CLINICAL TRIAL: NCT04799548
Title: A Phase II Study of Neoadjuvant Transcatheter Arterial Chemoembolization（TACE）Plus PD-1 Antibody (Tislelizumab) in the Locally Advanced Stomach Adenocarcinoma
Brief Title: A Phase II Study of TACE Plus PD-1 Antibody in the Locally Advanced Stomach Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSGC-TACiE04
Record Dates: First submitted 2021-01-31; First posted 2021-03-16 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Advanced Gastric Cancer
Keywords: Stomach Cancer; transcatheter arterial chemoembolization; PD-1; PD-L1; neoadjuvant therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant TACE plus Tislelizumab (Experimental)
  Interventions: Drug: Transcatheter Arterial Chemoembolization; Drug: Tislelizumab

INTERVENTIONS:
Drug: Transcatheter Arterial Chemoembolization — Patients will sequentially receive one cycle TACE (3 weeks), one cycle SOX regimen (3 weeks), one cycle TACE (3 weeks) and one cycle SOX (3 weeks) regimen, a total of 12-week neoadjuvant therapy.
  TACE cycle: Day 1: trans-femorally performed with infusion of oxaliplatin (85 mg/m2) into tumor blood vessels. Then, Embosphere® Microspheres (300-500 μm) will be injected for embolism. Day 1-14: Oral Tegafur Gimeracil Oteracil Potassium Capsule 40-60 mg bid.
  SOX cycle: Day 1: Oxaliplatin 130mg/m2 intravenous. Day 1-14: Oral Tegafur gimeracil oteracil potassium capsule 40-60 mg bid.
Drug: Tislelizumab — PD-1 antibody Tislelizumab will be administrated by 200mg, ivgtt, q3w throughout 12-week neoadjuvant treatment.

SUMMARY:
This study is a phase II, prospective, single-center, single-arm trial to evaluate the efficacy and safety of the combination of neoadjuvant transcatheter arterial chemoembolization (TACE) and PD-1 antibody Tislelizumab in the locally advanced stomach adenocarcinoma. The primary purpose of this study is to evaluate the pathologic complete response (pCR) rate of TACE plus Tislelizumab. The second purpose is to evaluate pathologic response rate (pRR), objective Response Rate (ORR), overall survival (OS) and progression-free survival (PFS) of the patients enrolled in this study.

DETAILED DESCRIPTION:
The treatment of advanced gastric cancer has been a significant global health problem. With surgery still the backbone, various clinical trials have shown the benefit of perioperative treatment to gastric cancer patients.

The report of transcatheter arterial chemoembolization (TACE) treatment in gastric cancer is relatively limited, though different case reports have showed its efficacy and safety in advanced gastric cancer. With transarterial infusion chemotherapy, TACE increases the local concentration of chemotherapeutic agents and reduces adverse reaction. With embolization, TACE blocks the blood supply and causes the necrosis of tumors, in this way exposing tumor antigen and promoting tumor immunity. The combination of TACE and PD-1 antibody is expected to further boost tumor immunity.

Meanwhile, Noman et.al. reported hypoxia could upregulate PD-L1 by activating HIF-1alpha. So, embolism may lead to immune evasion of tumors by upregulating PD-L1, but on the other side generate targets for PD-1/PD-L1 therapies.

Based on those knowledges, we designed this phase II, prospective, single-center, single-arm trial to evaluate the efficacy and safety of the combination of neoadjuvant transcatheter arterial chemoembolization (TACE) and PD-1 antibody Tislelizumab in the locally advanced stomach adenocarcinoma. The primary purpose of this study is to evaluate the pathologic complete response (pCR) rate of TACE plus Tislelizumab. The second purpose is to evaluate pathologic response rate (pRR), objective Response Rate (ORR), overall survival (OS) and PFS (progression-free survival) of the patients enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 75 years old;
2. KPS score >=80;
3. Gastric adenocarcinoma diagnosed pathologically;
4. According to endoscopic ultrasonography/enhanced CT/MRI/PET-CT examination and laparoscopic exploration, clinical staging is determined to be cT3/4aN+M0 (according to AJCC TNM 8th edition);
5. According to the RECIST1.1 standard, there is at least one evaluable lesion in the abdominal CT/MRI;
6. The surgeons participating in this study judged the lesion to be resectable;
7. Physical condition allows the surgery;
8. The blood routine and biochemical indexes of the subjects met standards within 7 days before enrollment:
9. There are no serious concomitant diseases that make the survival time <5 years;
10. Female subjects with fertility are not allowed to get pregnant or breastfeeding;
11. Be willing and able to comply with the plan and follow-up procedures during the research period.

Exclusion Criteria:

1. There are any signs of distant metastasis or local unresectable factors;
2. Those who are allergic to contrast agents;
3. Those who have received cytotoxic chemotherapy, radiotherapy, immunotherapy or radical surgery for the treatment of this gastric cancer, except for corticosteroids;
4. Patients who have active autoimmune diseases or have a history of autoimmune diseases but may relapse;
5. Any active malignant tumors within 2 years, except the specific cancers under study in this trial and locally recurring cancers that have been cured (such as resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast cancer);
6. There is uncontrollable pleural effusion, pericardial effusion or ascites that requires frequent drainage within 14 days before enrollment;
7. Patients with gastrointestinal bleeding within two weeks prior to enrollment, or those with high bleeding risk as judged by the investigators;
8. Gastrointestinal perforation and/or fistula occurred within 6 months before enrollment;
9. Upper gastrointestinal obstruction or abnormal physiological function or suffering from malabsorption syndrome, which may affect the absorption of drugs;
10. Weight loss >=20% within 2 months before enrollment;
11. A history of the following lung diseases: interstitial lung disease, non-infectious pneumonia, pulmonary fibrosis, acute lung disease, etc.;
12. There are uncontrollable systemic diseases including diabetes, hypertension, etc.;
13. Severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis, HIV infection, etc.;
14. Untreated patients with chronic hepatitis B or chronic HBV carriers with hepatitis B virus (HBV) DNA exceeding 500 IU/mL, or hepatitis C virus (HCV) RNA positive patients should be excluded;
15. Any of the following cardiovascular risk factors (refer to Research Guide)
16. Known peripheral nerve disease >=NCI CTCAE Grade 1. However, patients with only the disappearance of the deep tendon reflex (DTR) need not be excluded;
17. Moderate or severe renal damage [creatinine clearance equal to or lower than 50 ml/min (calculated according to the Cockroft and Gault equation)], or serum creatinine>ULN;
18. People with known dihydropyrimidine dehydrogenase (DPD) deficiency;
19. Those who are allergic to any research drug ingredients;
20. Have had allogeneic stem cell transplantation or organ transplantation;
21. Patients requiring systemic treatment with corticosteroids (dose higher than 10 mg/d of prednisone or equivalent doses of similar drugs) or other immunosuppressive agents <=14 days before enrollment.
22. Have received live vaccines within 4 weeks before enrollment. (Remarks: Seasonal flu vaccines are usually inactivated vaccines and are allowed to be used. Vaccines used in the nasal cavity are live vaccines and are not allowed.);
23. Have received immunotherapy (such as interleukin, interferon, thymosin, etc.) or any trial treatment within 28 days or 5 half-lives (whichever is shorter, but at least 14 days) before enrollment;
24. Palliative radiotherapy was performed within 14 days before enrollment;
25. Have received anti-PD-1, anti-PD-L1, anti-PD-L2 or any other specific targeting T cell costimulation or checkpoint pathway antibodies or drug therapy;
26. Underwent major surgery within 28 days prior to enrollment, unless the surgery was minimally invasive (for example, central venous catheterization via peripheral venipuncture [PICC]);
27. For people with a history of uncontrolled epilepsy, central nervous system disease, or mental disorder, the investigator will determine whether the clinical severity hinders the signing of informed consent or affects the patient's compliance with oral medications;
28. There is a potential medical condition or alcohol/drug abuse or dependence that the investigator believes is not conducive to the administration of the study drug or that affects the interpretation of drug toxicity or adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response (pCR) rate | 1 months

SECONDARY OUTCOMES:
pathologic response rate (pRR) | 1 months
objective Response Rate (ORR) | 1 months
overall survival (OS) | 3 years
progression-free survival (PFS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xuefei Wang, MD, phD, Principal Investigator — Fudan University
Locations (1):
- ZhongShan hospital Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scharping NE, Menk AV, Whetstone RD, Zeng X, Delgoffe GM. Efficacy of PD-1 Blockade Is Potentiated by Metformin-Induced Reduction of Tumor Hypoxia. Cancer Immunol Res. 2017 Jan;5(1):9-16. doi: 10.1158/2326-6066.CIR-16-0103. Epub 2016 Dec 9. PMID 27941003
- [Background] Su Z, Shu K, Kang M, Wang G. Pathological complete response from oral chemotherapy combined with trans-arterial chemotherapy and embolization in an unresectable gastric cancer patient: A case report. Medicine (Baltimore). 2019 Jun;98(25):e16075. doi: 10.1097/MD.0000000000016075. PMID 31232946
- [Background] Wu ZF, Cao QH, Wu XY, Chen C, Xu Z, Li WS, Yao XQ, Liu FK. Regional Arterial Infusion Chemotherapy improves the Pathological Response rate for advanced gastric cancer with Short-term Neoadjuvant Chemotherapy. Sci Rep. 2015 Dec 1;5:17516. doi: 10.1038/srep17516. PMID 26620627
- [Background] Zhang CW, Zou SC, Shi D, Zhao DJ. Clinical significance of preoperative regional intra-arterial infusion chemotherapy for advanced gastric cancer. World J Gastroenterol. 2004 Oct 15;10(20):3070-2. doi: 10.3748/wjg.v10.i20.3070. PMID 15378797
- [Background] Friedlander M, Meniawy T, Markman B, Mileshkin L, Harnett P, Millward M, Lundy J, Freimund A, Norris C, Mu S, Wu J, Paton V, Gao B. Pamiparib in combination with tislelizumab in patients with advanced solid tumours: results from the dose-escalation stage of a multicentre, open-label, phase 1a/b trial. Lancet Oncol. 2019 Sep;20(9):1306-1315. doi: 10.1016/S1470-2045(19)30396-1. Epub 2019 Aug 1. PMID 31378459
- [Background] Xu J, Bai Y, Xu N, Li E, Wang B, Wang J, Li X, Wang X, Yuan X. Tislelizumab Plus Chemotherapy as First-line Treatment for Advanced Esophageal Squamous Cell Carcinoma and Gastric/Gastroesophageal Junction Adenocarcinoma. Clin Cancer Res. 2020 Sep 1;26(17):4542-4550. doi: 10.1158/1078-0432.CCR-19-3561. Epub 2020 Jun 19. PMID 32561664